CLINICAL TRIAL: NCT07341464
Title: Acceptability (Including Gastrointestinal Tolerance and Compliance) of a Paediatric and Adult Bolus Tube Feed With Food Blends
Brief Title: Acceptability and Tolerance Study of Bolus Tube Feed With Food Blends
Acronym: Blends
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BTB 001; IRAS ID 341165 (Other: West of Scotland REC 5 West of Scotland Research Ethics Service, Ward 11, Dykebar Hospital Grahamston Road PAISLEY PA2)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Oncology
MeSH Terms: conditions — Cerebral Palsy; Neoplasms | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptability and Tolerance Study of bolus tube feed with food blends (Other): Arm one will act as their own controls
  Interventions: Dietary Supplement: Tube feed

INTERVENTIONS:
Dietary Supplement: Tube feed — Dose intake and duration.

SUMMARY:
This is a prospective acceptability study to evaluate the gastrointestinal tolerance and compliance of a bolus tube feed over a 28 -day period for up to 50 participants.

The enteral bolus formula is for the dietary management of patients with short bowel syndrome; intractable malabsorption; preoperative preparation of undernourished patients; inflammatory bowel disease; total gastrectomy; dysphagia; bowel fistulae; feeding intolerances, developmental disabilities, and disease related malnutrition.

DETAILED DESCRIPTION:
The study will collect data in 50 children and adults over a period of 28 days. Gastrointestinal tolerance will be collected over 7 days and formula intake will be over 28 days. A patient satisfaction questionnaire will be completed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 1 -15 years for children and 15 years and above for adults of requiring 1 or more bolus tube feed alongside their usual tube feed or home-made blended diet as part of their dietary management for disease related malnutrition.
* Patients well-established and stable on current enteral tube feed or home-made blended diet.
* Gastrostomy fed only.
* Willingly given, written, informed consent from patient/caregiver

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator.
* Under 1 years of age
* Patients who have a nasogastric and jejunal feeding tubes
* Patients on total parenteral nutrition
* Known food allergies to any ingredients listed in appendix 1.
* Patients with significant renal or hepatic impairment
* Participation in another interventional study within 2 weeks of this study.
* Patients with known or suspected ileus or mechanical bowel obstruction

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Measure of Gastrointestinal tolerance | 7 days
  Severity of symptoms such as reflux, vomiting, constipation, diarrhoea as a four-point likert scale (none, mild, moderate, severe).
Daily record of formula intake. | 28 days
  Measure of formula intake in mL.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Queen Medical Hospital Nutrition and Dietetics, Nottingham
  - Dietetic Team 1st floor Kings Court 1, Charles Hastings Way,, Worcester

IPD SHARING:
Plan to Share IPD: No